CLINICAL TRIAL: NCT07216469
Title: Myocardial Stiffness in Amyloidosis by Magnetic Resonance Elastography - AMREloid Study
Brief Title: A Study Of Myocardial Stiffness In Amyloidosis With Magnetic Resonance Elastography
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ian C. Chang, Principal Investigator, Mayo Clinic
Other Study IDs: 25-006581
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Amyloidosis
  Interventions: Diagnostic Test: Magnetic Resonance Elastography (MRE)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Elastography (MRE) — Patients will undergo a cardiac MRI with the addition of continuous free-breathing and breath-held MRE sequences.

SUMMARY:
This is a prospective case control study to determine the feasibility and utility of myocardial stiffness assessment by cardiac magnetic resonance elastography (MRE) in patients with cardiac amyloidosis.

ELIGIBILITY:
Inclusion Criteria

Subjects are eligible to be included in the study if all the following criteria apply:

1. Adult, age 20 and greater
2. Subject is clinically stable without cardiovascular-related hospitalizations within 2 weeks prior to enrollment as assessed by the investigators
3. Subject is able to provide written informed consent and is willing and able to complete study procedures
4. Subject must meet criteria for either ATTR cardiac amyloidosis or AL cardiac amyloidosis from review of medical records as specified below:

   a. ATTR cardiac amyloidosis based on meeting all the following criteria:

   i. Diagnosis of amyloidosis within ten years prior to study screening

   ii. Transthyretin amyloid deposits in cardiac tissue OR Technetium (99mTc) bone scintigraphy with grade 2 or 3 cardiac uptake OR Transthyretin amyloid deposits in non-cardiac tissue with echocardiographic evidence of cardiac involvement or an end-diastolic mean wall thickness > 12 mm OR Transthyretin amyloid deposits in non-cardiac tissue with cardiac MRI diagnostic of amyloidosis OR Clinical diagnosis of cardiac amyloidosis by the clinical provider

   b. AL cardiac amyloidosis based on meeting all the following criteria:

   i. Diagnosis of amyloidosis within ten years prior to study screening

   ii. Histopathologic diagnosis of amyloidosis with AL protein identification

   iii. Cardiac involvement as defined by: Amyloid deposits in cardiac deposits OR Echocardiography with an end-diastolic mean wall thickness > 12 mm in the absence of other causes OR Elevated NT-proBNP (>332 ng/L) in the absence of renal failure or atrial fibrillation OR Cardiac MRI diagnostic of amyloidosis OR Clinical diagnosis of cardiac amyloidosis by the clinical provider

   Exclusion Criteria

   Patients are ineligible to be included in the study if any of the following criteria apply:

1. Unable to consent or unable to complete all study procedures 2. Unable to ambulate for 6 minutes (confirmed at study coordinator visit) 3. Unable to maintain in supine position for 30 minutes 4. Unable to maintain breath-holding for 10 seconds (confirmed at study coordinator visit) 5. Contraindications for safe MRI scanning (e.g., uncontrolled claustrophobia, cochlear implant, implanted neural stimulator) 6. Presence of implantable cardiac pacemaker or defibrillator 7. History of complex congenital heart disease, prosthetic valves, prosthesis in the main pulmonary artery or ascending thoracic aorta 8. Significant artifact from prior MRI studies 9. Pregnant or breast-feeding women 10. Weight equal to or greater than 155 kg 11. In the judgment of the investigator, has clinically relevant ongoing medical condition or laboratory abnormalities or other condition that might jeopardize the participants safety, increase the participants risk from participation, interfere with the study, or confirmed study results

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Mayo Clinic's Cardiology, Hematology, and Cardiovascular Imaging clinics."
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects able to complete a Magnetic Resonance Elastography exam | Baseline
  Magnetic Resonance Elastography exam completion will be determined by signal to noise (SNR) ratio
Mean Myocardial Stiffness | Baseline
  Mean Myocardial stiffness will be measured by magnetic resonance elastography during early systole, end systole, early diastole and end diastole (kPa).

CONTACTS AND LOCATIONS:
Overall Officials: Ian Chang, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No